CLINICAL TRIAL: NCT06892795
Title: Construction of a Risk Prediction Model for Hypothermia During Surgery in Pediatric Under General Anesthesia Based on Machine Learning Algorithm
Brief Title: Constructing a Risk Prediction Model for Intraoperative Hypothermia in Children Under General Anesthesia
Status: Enrolling by invitation | Type: Observational
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Huanglu Lan, Principal Investigator, Harbin Medical University
Other Study IDs: LC2024-141; YJSCX2024-124HYD (Other Grant/Funding Number: Harbin Medical University)
Record Dates: First submitted 2025-03-05; First posted 2025-03-25 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Hypothermia, Accidental; Hypothermia; Anesthesia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — The investigators will not collect any biological specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hypothermia: Core body temperature below 36°C during surgery
- Non-hypothermia: Core body temperature ≥ 36°C during surgery

SUMMARY:
Intraoperative hypothermia refers to a core body temperature below 36.0°C during surgery, which is common in surgical patients. Due to the fact that children's body temperature regulation function is not yet fully developed, they are light in weight, and their blood vessels are superficial, children are very susceptible to the influence of environmental temperature. With the effects of anesthetic drugs, exposure of the surgical field, and disinfection of the surgical area, children face a higher risk of intraoperative hypothermia than adult patients. Studies have shown that the incidence of intraoperative hypothermia can be as high as 80%. Intraoperative hypothermia can lead to increased adverse cardiovascular events, poor coagulation, slower healing of surgical incisions, or wound infection, threatening the health of children, resulting in prolonged postoperative hospitalization and increased hospitalization costs. Therefore, there is an urgent need to develop a tool for predicting intraoperative hypothermia suitable for children, identify high-risk groups early, and take preventive measures as soon as possible, thereby reducing a series of complications caused by hypothermia. The purpose of this study is to clarify the current status and risk factors affecting intraoperative hypothermia in children, to provide a theoretical basis for clinical medical staff to provide intraoperative thermal insulation care for children, and on this basis to construct an intraoperative hypothermia risk prediction model to identify the probability of hypothermia in children at an early stage, so as to take targeted thermal insulation measures.

DETAILED DESCRIPTION:
The study first clarified the overall incidence and influencing factors of IOH in children through meta-analysis, combined with expert consultation to determine potential predictive variables, and developed a data questionnaire for this study. The second part of the study will collect data prospectively, use four algorithms in machine learning, including logistic regression, decision tree, random forest, and support vector machine, to build an excellent intraoperative hypothermia risk prediction model, and conduct internal verification of the model. The third part of the study prospectively collects sample data to complete external verification of time period and space. The constructed model still has good predictive ability in the new data set. Finally, some models are visualized to form intuitive and easy-to-understand charts or interfaces.

ELIGIBILITY:
Inclusion Criteria:

* Age < 16 years old;
* Anesthesia includes general anesthesia;
* Anesthesia duration > 30 minutes.

Exclusion Criteria:

* Cardiac surgery or other procedures that require lowering the child's body temperature;
* Refusing to participate in this study;
* ASA grade >Ⅳ;
* Abnormal basal body temperature, preoperative core body temperature <36.0℃ or >38.0℃;
* Hyperthyroidism or hypothyroidism and other diseases that affect body temperature;
* The core body temperature cannot be measured due to surgery or ear canal disease.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric surgical patients receiving general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 562 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Core body temperature | The investigators will measure the child's core body temperature when the child enters the operating room, after induction of anesthesia, and then every 30 minutes until the end of the operation.
  Use an infrared electronic ear thermometer to measure the child's eardrum temperature as the core body temperature.

CONTACTS AND LOCATIONS:
Overall Officials: Huanglu Lan, Principal Investigator — The Sixth Affiliated Hospital of Harbin Medical University
Locations (1):
- The Sixth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided